CLINICAL TRIAL: NCT01321476
Title: Contribution of Hepatic and Intestinal Lipoproteins to Human Atherosclerosis
Acronym: Carotid
Status: Withdrawn | Type: Observational
Why Stopped: Study was never initiated and internal decision to discontinue initiation process
Sponsor: Piedmont Healthcare (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Joseph Miller, MD, Piedmont Heart Institute
Other Study IDs: Carotid
Record Dates: First submitted 2011-03-14; First posted 2011-03-23 (Estimated); Last update posted 2013-09-05 (Estimated); Status verified 2011-07

CONDITIONS: Heart Disease
MeSH Terms: conditions — Heart Diseases

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Carotid artery tissue Liver biopsy tissue Intestinal biopsy tissue Cell cultures
Oversight: Data Monitoring Committee: No

SUMMARY:
This study will use excess tissue from endoscopic or surgical procedures to examine the elements of plaque that are found in the carotid walls of patients who have a type of heart and blood vessel disease called atherosclerosis. Tissue will be collected from patients undergoing carotid procedures as well as patients undergoing liver and/or intestinal biopsies. This lab study will examine the different types of proteins that play a role in developing heart plaque.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Scheduled for a clinically indicated, standard-of-care carotid endarterectomy (CEA) OR scheduled for a clinically indicated, standard-of- care surgical, laparoscopic or endoscopic intestinal biopsy or excision OR scheduled for a clinically indicated, standard-of-care surgical, laparoscopic or endoscopic liver biopsy or partial resection/excision
* Ability and willingness to consent and Authorization for use of PHI

Exclusion Criteria:

* Age ≤18 years
* Inability or unwillingness to consent and Authorization for use of PHI
* FOR CAROTID PATIENTS - history of carotid trauma, that is determined by the Principal Investigator to significantly have changed the carotid tissue structure
* FOR CAROTID PATIENTS - history of middle- or large-vessel vasculitis, that is determined by the Principal Investigator to significantly have changed the carotid tissue structure

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients undergoing a carotid, liver, and/or intestinal biopsy
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)

PRIMARY OUTCOMES:
Demonstrated Plaques | up to 30 months
  Presence of both liver and intestinally derived lipoprotein particles demonstrated in human atherosclerotic plaques.

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Miller, MD, Principal Investigator — Piedmont Heart Institute/Piedmont Hospital